CLINICAL TRIAL: NCT04196231
Title: Durability of Combination of Insulin and GLP-1 Receptor Agonist or SGLT-2 Inhibitors Versus Basal Bolus Insulin Regimen in Type 2 Diabetes: a Randomized Controlled Trial
Brief Title: Durability of Combination of Insulin and GLP-1 Receptor Agonist or SGLT-2 Inhibitors Versus Basal Bolus Insulin Regimen in Type 2 Diabetes (BEYOND)
Acronym: BEYOND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Katherine Esposito, Full Professor of Endocrinology and Metabolic Diseases, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEYOND Protocol
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; GLP-1RA; SGLT-2i; basal insulin; basal bolus; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira; Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FR insulin/GLP-1RA (Active Comparator): Patients in this arm will receive one of these fixed ratio combo of insulin and GLP-1RAs, according to the current clinical practice and the drugs' data sheet: IDegLira or IGlarLixi
  Interventions: Drug: IDegLira; Drug: IGlarLixi
- Insulin/SGLT-2i (Active Comparator): Patients in this arm will receive the basal insulin used before the randomization and one of these SGLT-2i according to the current clinical practice and the drugs' data sheet: canagliflozin, dapagliflozin or empagliflozin.
  Interventions: Drug: Insulin/Canaglifozin; Drug: Insulin/Dapaglifozin; Drug: Insulin/Empaglifozin
- Basal Bolus (Active Comparator): Patients in this arm will receive a basal insulin (glargine, glargine-300 or degludec) at bed-time plus 3 injections of a short-acting insulin analogue (aspart, lispro or glulisine) before meals
  Interventions: Drug: Basal Bolus

INTERVENTIONS:
Drug: IDegLira — IDegLira will be started at 16 dose steps (16 U insulin degludec plus 0.58 mg liraglutide, once daily). On the basis of prebreakfast self-monitored blood glucose measurements doses of IDegLira will be titrated individually twice per week to achieve a prebreakfast plasma glucose of 80-130 mg/dL by use of an algorithm (adding 2 dose steps for prebreakfast plasma glucose >130 mg/dL; no dose change for prebreakfast plasma glucose of 80-130 mg/dL; reducing 2 dose steps for prebreakfast plasma glucose < 80 mg/dL). The daily dose of IDegLira could be titrated to 50 dose steps (50 U insulin degludec plus 1.8 mg liraglutide).
  Arms: FR insulin/GLP-1RA
Drug: IGlarLixi — IGlarLixi will be started at 10 dose steps (10 U insulin glargine plus 5 mcg lixisenatide, once daily). On the basis of prebreakfast self-monitored blood glucose measurements, doses of IGlarLixi will be titrated individually once per week to achieve a prebreakfast plasma glucose of 80-130 mg/dL by use of an algorithm (adding 2 dose steps for prebreakfast plasma glucose >130 mg/dL; no dose change for prebreakfast plasma glucose of 80-130 mg/dL; reducing 2 dose steps for prebreakfast plasma glucose < 80 mg/dL). The daily dose of IGlarLixi could be titrated to 60 dose steps (60 U insulin degludec plus 20 mcg lixisenatide).
  Arms: FR insulin/GLP-1RA
Drug: Insulin/Canaglifozin — Patients in this arm will continue the basal insulin used before the randomization, with dosage titration on the basis of the following algorithm: adding 2 units for prebreakfast plasma glucose >130 mg/dL; no dose change for prebreakfast plasma glucose of 80-130 mg/dL; reducing 2 units for prebreakfast plasma glucose < 80 mg/dL. Moreover, they will be assigned to canaglifozin, according to the current clinical practice and the drugs' data sheet. Canagliflozin will be started at 100 mg daily per oral administration, and augmented to 300 mg/per day if required (HbA1c >7.5 after 12 weeks).
  Arms: Insulin/SGLT-2i
Drug: Insulin/Dapaglifozin — Patients in this arm will continue the basal insulin used before the randomization, with dosage titration on the basis of the following algorithm: adding 2 units for prebreakfast plasma glucose >130 mg/dL; no dose change for prebreakfast plasma glucose of 80-130 mg/dL; reducing 2 units for prebreakfast plasma glucose < 80 mg/dL. Moreover, they will be assigned to dapaglifozin, according to the current clinical practice and the drugs' data sheet. Dapagliflozin will be started at 10 mg daily per oral administration
  Arms: Insulin/SGLT-2i
Drug: Insulin/Empaglifozin — Patients in this arm will continue the basal insulin used before the randomization, with dosage titration on the basis of the following algorithm: adding 2 units for prebreakfast plasma glucose >130 mg/dL; no dose change for prebreakfast plasma glucose of 80-130 mg/dL; reducing 2 units for prebreakfast plasma glucose < 80 mg/dL. Moreover, they will be assigned to empaglifozin, according to the current clinical practice and the drugs' data sheet. Empagliflozin will be started at 10 mg daily per oral administration, and augmented to 25 mg/per day if required (HbA1c >7.5 after 12 weeks).
  Arms: Insulin/SGLT-2i
Drug: Basal Bolus — Patients in this arm will continue the basal insulin (glargine, degludec or glargine-300) used before the randomization. The insulin titration will be guided by the medical staff, according to the following algorithm: adding 2 units of basal insulin for prebreakfast plasma glucose >130 mg/dL; no dose change for prebreakfast plasma glucose of 80-130 mg/dL; reducing 2 units of basal insulin for prebreakfast plasma glucose < 80 mg/dL. The short acting insulin analogue (lispro, aspart or glulisine) will be started at the dosage of 4 units before meals (3 times per day) and will be titrated twice a week until achieving pre-prandial glucose values ranging from 80-130 mg/dL.
  Arms: Basal Bolus

SUMMARY:
BEYOND represents an open-label, parallel, three-arm randomized controlled trial, aimed at evaluating the effects of combination therapy of fixed ratio basal insulin/GLP-1 receptor agonist (GLP-1RA) or basal insulin/SGLT-2 inhibitors (SGLT-2i) on the durability of the glycemic control, as compared with the basal bolus insulin regimen, in people with type 2 diabetes failing to achieve glycemic targets with injective therapy. The potential benefits for participants in the study include the possibility of improving the glyco-metabolic control with drugs that have been evaluated as safe and protective for the heart and the kidneys. The primary outcome of the study is the mean HbA1c change between groups at six months. Participants in the study will be followed for subsequent 18 months in order to evaluate the durability of glycemic control and the chenge of other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Poor glycemic control (HbA1c ≥7.5%)
* Stable basal bolus insulin regimen for almost a year, eventually associated with metformin.

Exclusion Criteria:

* Type 1 diabetes or secondary diabetes;
* Previous treatment for the last three months with GLP-1RA or DPP-4 inhibitors;
* Hypersensitivity towards active substances or other ingredients of the drugs used in the study
* Participation in other trial with experimental drugs within 30 days
* Diseases that represent contraindication to GLP-1RA use (pancreatitis, gallstones)
* Pregnancy or planned pregnancy within the time of the study
* Serum creatinine > 1,3 mg/dL in women and >1,4 mg/dL in men
* eGFR < 30 mL/min
* Previous cancer or antineoplastic therapy for five years before randomization
* Current therapy with glucocorticoid (oral, topic or sistemic administration) or with antypsichotic drugs
* Previous ketoacidosis
* Any clinical, psychologic or psychiatric condition that is incompatible with the study according to the investigator

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Hba1c change | 6 months, 9 months, 12 months
  HbA1c group difference at 6 months
Proportions of patients with significant HbA1c change | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months
  Proportions of patients undergoing a reduction equal or higher than 0.5% as compared with baseline levels during the follow up

SECONDARY OUTCOMES:
Weight Change | Baseline, 6 months, 18 months
BMI Change | Baseline, 6 months, 18 months
Waist circumference change | Baseline, 6 months, 18 months
Blood pressure change | Baseline, 6 months, 18 months
Fasting glycemia change | Baseline, 6 months, 18 months
Post-prandial glycemia change | Baseline, 6 months, 18 months
C-peptide change | Baseline, 6 months, 18 months
Change in total daily insulin dose | Baseline, 6 months, 18 months
Change in lipide profile | Baseline, 6 months, 18 months
  Difference between groups in total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides
Change in eGFR | Baseline, 6 months, 18 months
Diabetes treatment satisfaction | Baseline, 6 months, 18 months
  In order to measure satisfaction with diabetes treatment regimens, we used the self-reported Diabetes Treatment Satisfaction Questionnaire. This instrument aims to assess levels of satisfaction in subjects using different treatment strategies. The questionnaire consists of eight questions: six questions addresses general satisfaction with a score from 0 to 6 for each question (0 = worst), that has to be computed in a total score ranging from 0 (=worst) to 36 (=best); among the remaining two questions, which has to be computed separately as two subscales, one concerns the perception of hyperglycemic events and another the perception of hypoglycemic events, both with a score from 0 (none of the time) to 6 (most of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Esposito, MD, PhD, Principal Investigator — Unit of Diabetology University of Campania Luigi Vanvitelli; Dario Giugliano, MD, Principal Investigator — Unit of Endocrinology and Metabolic Diseases University of Campania Luigi Vanvitelli; Giuseppe Bellastella, MD, PhD, Study Chair — Unit of Endocrinology and Metabolic Diseases University of Campania Luigi Vanvitelli; Maria Ida Maiorino, MD, PhD, Study Chair — Unit of Diabetology University of Campania Luigi Vanvitelli
Locations (1):
- Unit of Endocrinology and Metabolic Diseases, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giugliano D, Bellastella G, Maiorino MI, Esposito K. Beyond basal-bolus insulin regimen: Is it still the ultimate chance for therapy in diabetes? Diabetes Res Clin Pract. 2019 Nov;157:107922. doi: 10.1016/j.diabres.2019.107922. Epub 2019 Nov 9. No abstract available. PMID 31715201
- [Derived] Giugliano D, Longo M, Scappaticcio L, Caruso P, Gicchino M, Petrizzo M, Bellastella G, Maiorino MI, Esposito K. BEYOND 2 years: durability of metabolic benefits by simplification of complex insulin regimens in type 2 diabetes. Endocrine. 2024 Feb;83(2):399-404. doi: 10.1007/s12020-023-03547-9. Epub 2023 Oct 3. PMID 37787888
- [Derived] Giugliano D, Longo M, Caruso P, Di Fraia R, Scappaticcio L, Gicchino M, Petrizzo M, Bellastella G, Maiorino MI, Esposito K. Feasibility of Simplification From a Basal-Bolus Insulin Regimen to a Fixed-Ratio Formulation of Basal Insulin Plus a GLP-1RA or to Basal Insulin Plus an SGLT2 Inhibitor: BEYOND, a Randomized, Pragmatic Trial. Diabetes Care. 2021 Jun;44(6):1353-1360. doi: 10.2337/dc20-2623. Epub 2021 Apr 21. PMID 33883195